CLINICAL TRIAL: NCT05208229
Title: The Role of WB-MRI in the Evaluation of Prostate Cancer Patients Treated With Lu-PSMA
Brief Title: The Role of WB-MRI in the Evaluation of Prostate Cancer Patients Treated With Lutetium - Prostate Specific Membrane Antigen (Lu-PSMA)
Acronym: WB-LuPSMA
Status: Terminated | Type: Observational
Why Stopped: The study was linked to another protocol that is over
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: IRST185.08
Record Dates: First submitted 2021-02-25; First posted 2022-01-26 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Metastatic Castration Resistant Prostate Cancer (mCRPC)
Keywords: WB-MRI (Whole Body- Magnetic Resonance Imaging); 177Lu-PSMA 617; metastatic Castration Resistant Prostate Cancer (mCRPC); Radio Metabolic Therapy (RMT)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with mCRPC enrolled in the Tumor Institute of Romagna (IRST) 185.03 Lu-PSMA protocol: Patients with mCRPC enrolled in the IRST 185.03 Lu-PSMA study, performing baseline CT and WB-MRI examinations and at least one CT and WB-MRI re-evaluation.
  Interventions: Diagnostic Test: WB-MRI

INTERVENTIONS:
Diagnostic Test: WB-MRI — Baseline CT scan (minimum thorax/abdomen/pelvis) and WB-MRI evaluations will be collected: as per clinical practice and Tumor Institute of Romagna (IRST) 185.03 Lu-PSMA protocol, the assessments must not be performed more than 12 weeks prior to study entry and baseline WB-MRI should be performed within 2 weeks from CT scan; CT and WB-MRI will be done at the end of Lutetium 177 PSMA (177Lu-PSMA) therapy and during post-treatment follow-up

SUMMARY:
The role of WB-MRI in the evaluation of prostate cancer patients treated with Lu-PSMA

DETAILED DESCRIPTION:
Multicentric, observational, single arm, prospective, study.

All patients will undergo imaging assessments according to clinical practice or to Lu-PSMA Tumor Institute of Romagna (IRST) 185.03 protocol, as follows:

* Baseline, before the treatment with Lu-PSMA, CT and WB-MRI will be performed
* At the end of treatment with Lu-PSMA, CT and WB-MRI will be performed
* In post-treatment follow-up every 4 months, until progression or for 1 year, CT and WB-MRI will be performed.

Patients participating in this observational study will not be subjected to any additional procedure that falls outside the clinical practice or the study 185.03 Lu-PSMA trial at IRST.

ELIGIBILITY:
Inclusion Criteria:

- Patients with mCRPC enrolled in the Tumor Institute of Romagna (IRST) 185.03 Lu-PSMA protocol, performing baseline CT and WB-MRI examinations and at least one CT and WB-MRI re-evaluation.

Exclusion Criteria:

* no exclusion criteria

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with mCRPC enrolled in the IRST185.03 Lu-PSMA study
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-03-08 (Actual); Study Completion 2022-03-08 (Actual)

PRIMARY OUTCOMES:
disease progression | up to 42 months
  To evaluate whether WB-MRI allows earlier identification of disease progression in comparison to CT in mCRPC patients based on imaging criteria.

SECONDARY OUTCOMES:
Reproducibility of The Metastasis (MET) Reporting And Data System (RADS) for Prostate Cancer (P) (MET - RADS - P) assessment of WB-MRI | up to 42 months
  To assess reproducibility of MET-RADS-P assessment of WB-MRI in metastatic prostate disease. The reproducibility of MET-RADS-P assessment of WB-MRI in metastatic prostate disease will be assessed using the concordance of the Response Assessment Categories (RAC) scores (RACs) assigned by two independent observers.
response with WB-MRI compared to other assessment | up to 42 months
  Quantitative metrics describing patterns of response that can be observed on WB-MRI, on CT, and possibly on Ga PSMA Positron Emission Tomography (PET)/CT.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Paganelli, MD, Study Chair — IRST IRCCS
Locations (2):
- Italy (2):
  - IRCCS Istituto Romagnolo per lo Studio dei Tumori "Dino Amadori" - IRST s.r.l., Meldola, Forlì-Cesena
  - European Institute of Oncology, Milan